CLINICAL TRIAL: NCT04072549
Title: Reducing Health Disparities in Childhood Obesity Using Financial Incentives in Low-income Households
Brief Title: Reducing Health Disparities in Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Michael Beets, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00086238
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: We will compare changes in weight status and obesogenic behaviors of children from low-income households randomized to one of two conditions: free summer programming or comparison/control.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Summer Programming (Experimental): The summer day camps are not singularly focused, such as sport camps or academic only camps. Rather, the camps provide indoor and outdoor opportunities for children to be physically active each day, provide enrichment and academic programming, as well as provide breakfast, lunch, and snacks. To standardize programming, the schools operate their camps on the same daily schedules which are developed by the same district-level personnel, with identical programmatic content delivered across all schools. The schools also provide the same meals to all children enrolled. The meals adhere to the Summer Food Service Program nutrition guidelines and are reimbursed through existing federal food programs.
  Interventions: Behavioral: Free Summer Programming
- Comparison/Control (No Intervention): The children in the control group will be children enrolled in the same schools as those randomized to receive summer programming. The comparison/control group will not receive a voucher to attend a summer camp.

INTERVENTIONS:
Behavioral: Free Summer Programming — The summer day camps are not singularly focused, such as sport camps or academic only camps. Rather, the camps provide indoor and outdoor opportunities for children to be physically active each day, provide enrichment and academic programming, as well as provide breakfast, lunch, and snacks. To standardize programming, the schools operate their camps on the same daily schedules which are developed by the same district-level personnel, with identical programmatic content delivered across all schools. The schools also provide the same meals to all children enrolled. The meals adhere to the Summer Food Service Program nutrition guidelines and are reimbursed through existing federal food programs.
  Arms: Summer Programming

SUMMARY:
In this study, we will address cost barriers to participating in summer programs and hypothesize this will lead to marked improvements in children's obesogenic behaviors and a reduction in excessive, unhealthy weight gain over summer.

DETAILED DESCRIPTION:
For this study, we will rigorously test the impact of providing access to existing community-operated summer programs on weight status (i.e., BMI z-score) and obesogenic behaviors of 1st-3rd grade children from low-income households. Using a pragmatic, Type II hybrid effectiveness-implementation randomized design, we will compare changes in weight status and obesogenic behaviors of children from low-income households randomized to one of two conditions: free summer programming or comparison/control.

ELIGIBILITY:
Inclusion Criteria:

1st through 3rd grade students in the participating schools.

Exclusion Criteria:

The only exclusion criteria will be the diagnosis of an intellectual disability, such as:

Autism Spectrum Disorder Down Syndrome Fragile X Fetal Alcohol and/or a physical disability, such as wheelchair use

This decision was made because of the added resources required to evaluate these children, as well as the inability to sample enough of these children to adequately draw conclusions.

No other exclusion criteria will be used.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 651 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
BMI | Baseline and 3 months
  Change in Body Mass Index - height and weight

SECONDARY OUTCOMES:
Physical Activity | Baseline and 2 months
  Accelerometer-derived physical activity (minutes per day)
Sleep | Baseline and 2 months
  Accelerometer-derived sleep (minutes per day)
Diet | Baseline and 2 months
  Parent report of child dietary intake (healthy eating index)
Screen Time | Baseline and 2 months
  Parent report of screen time usage (minutes per day)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Carolina, Columbia, South Carolina
  - Michael Beets, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beets MW, Burkart S, Pfledderer CD, Adams E, Weaver RG, Armstrong B, Brazendale K, Zhu X, Chen B, McLain A. Impact of free summer day camp on physical activity behaviors and screentime of elementary-age children from low-income households: a randomized clinical trial. Int J Behav Nutr Phys Act. 2025 Dec 29;22(1):159. doi: 10.1186/s12966-025-01852-2. PMID 41466370
- [Derived] Beets MW, Burkart S, Pfledderer C, Adams E, Glenn Weaver R, Armstrong B, Brazendale K, Zhu X, Chen B, McLain A. Impact of Free Summer Day Camp on Physical Activity Behaviors and Screentime of Elementary-age Children from Low-Income Households: A Randomized Clinical Trial. Res Sq [Preprint]. 2025 May 13:rs.3.rs-6353093. doi: 10.21203/rs.3.rs-6353093/v1. PMID 40470250
- [Derived] Beets MW, Burkart S, Pfledderer C, Adams E, Weaver RG, Armstrong B, Brazendale K, Zhu X, Chen B, McLain A. Free Summer Programming and Body Mass Index Among Schoolchildren From Low-Income Households: A Randomized Clinical Trial. JAMA Pediatr. 2024 Dec 1;178(12):1252-1259. doi: 10.1001/jamapediatrics.2024.3693. PMID 39401051